CLINICAL TRIAL: NCT03171311
Title: European Trial on Optical Coherence Tomography Optimized Bifurcation Event Reduction - The OCTOBER Trial -
Brief Title: The OCTOBER Trial - European Trial on Optical Coherence Tomography Optimized Bifurcation Event Reduction (OCTOBER)
Acronym: OCTOBER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, phd, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-161-16
Record Dates: First submitted 2017-05-28; First posted 2017-05-31 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ischaemic Heart Disease; Ischemic Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia | interventions — Angioplasty, Balloon, Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiographic guided PCI (Active Comparator): Angiographic guided PCI is revascularization by percutaneous coronary intervention (PCI) and optional use of intravascular ultrasound (IVUS).
  Interventions: Procedure: Angiographic guided PCI
- OCT guided PCI (Experimental): OCT guided PCI is percutaneous coronary intervention (PCI) guided by systematic use of intravascular optical coherence tomography (OCT)
  Interventions: Procedure: OCT guided PCI

INTERVENTIONS:
Procedure: Angiographic guided PCI — Angiographic guided PCI is percutaneous coronary intervention performed by standard angiographic guided techniques
  Other Names: PCI, percutaneous transluminal coronary angioplasty (PTCA)
  Arms: Angiographic guided PCI
Procedure: OCT guided PCI — OCT guided PCI is percutaneous coronary intervention (PCI) guided by intra vascular optical coherence tomography (OCT) scans
  Other Names: OCT
  Arms: OCT guided PCI

SUMMARY:
The purpose is to compare median two-year clinical outcome after OCT guided vs. standard guided revascularization of patients requiring complex bifurcation stent implantation

DETAILED DESCRIPTION:
Coronary bifurcation lesions with stenosis in a large side branch may require complex stent implantation techniques with an elevated risk of suboptimal treatment results. Intra vascular optical coherence tomography (OCT) enables improved procedural control of correctable factors and may lead to optimized implantation results.

It is unknown if routine, systematic use of OCT scans during complex bifurcation stenting improves clinical outcome but present available evidence indicates advantages of OCT guidance that could translate into improved clinical outcome.

Hypothesis: Systematic OCT guided revascularization of patients with bifurcation lesions requiring complex stent implantation provides superior two-year clinical outcome compared to standard revascularization by PCI.

Methods: Investigator initiated and investigator sponsored, randomized (1:1), controlled, prospective, multicenter, superiority trial. Randomization is stratified for 1) Left main or non-Left main artery disease, and 2) up-front planned one-stent technique with kissing balloon inflation, or a two-stent technique.

Systematic OCT guidance is detailed for five complex stent implantation techniques. Standard treatment is angiographic based with optional use of intravascular ultrasound (IVUS).

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris, unstable angina pectoris, clinically stable non-STEMI.
* Age ≥18 yrs.
* Abel to provide written Informed consent and willing to comply with the specified follow-up contacts.

Angiographic inclusion criteria:

* Native coronary bifurcation de novo lesion
* More than 50% diameter stenosis in the main vessel (MV)
* More than 50% diameter stenosis in the side branch (SB) within 5 mm of the ostium.
* Reference size at least 2.75 mm in the main vessel (MV) and ≥2.5 mm in the SB.

Functional inclusion criteria:

Functional significance of the main vessel lesion or documented ischemia of the main vessel territory or other objective documentation of lesion significance. Objective evidence of ischemia is required for all treated lesions except for lesions with more than 80% diameter stenosis that may be considered significant.

Procedural inclusion criteria:

Indication for two-stent technique or one-stent technique with kissing balloon inflation

Exclusion Criteria:

* STEMI within 72 hours
* Cardiogenic shock
* Prior coronary artery bypass grafting (CABG) or planned CABG
* Renal failure with glomerular filtration rate (GFR) <50 mL/min per 1.73 m2
* Active bleeding or coagulopathy
* Life expectancy < 2 years
* Ejection fraction < 30%
* New York Heart Association (NYHA) class > II
* Relevant allergies (aspirin, clopidogrel, ticagrelor, contrast compounds, everolimus).

Angiographic exclusion criteria:

* Severe tortuosity around target bifurcation
* Chronic total occlusions
* Massive thrombus in Left main coronary artery
* Medina 0.0.1 lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1201 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of major adverse cardiac events (MACE) | 24 months
  Composite of cardiac death, target lesion myocardial infarction, ischaemic driven target lesion revascularization

SECONDARY OUTCOMES:
Study bifurcation oriented composite endpoint | 1 month
  Composite of cardiac death, target bifurcation myocardial infarction, target bifurcation revascularisation
Study bifurcation oriented composite endpoint | 12 months
  Composite of cardiac death, target bifurcation myocardial infarction, target bifurcation revascularisation
Study bifurcation oriented composite endpoint | 24 months
  Composite of cardiac death, target bifurcation myocardial infarction, target bifurcation revascularisation
Study bifurcation oriented composite endpoint | 36 months
  Composite of cardiac death, target bifurcation myocardial infarction, target bifurcation revascularisation
Study bifurcation oriented composite endpoint | 48 months
  Composite of cardiac death, target bifurcation myocardial infarction, target bifurcation revascularisation
Study bifurcation oriented composite endpoint | 60 months
  Composite of cardiac death, target bifurcation myocardial infarction, target bifurcation revascularisation
Patient oriented composite endpoint | 1 month
  Composite of all-cause mortality, myocardial infarction, any revascularisation, stroke
Patient oriented composite endpoint | 12 months
  Composite of all-cause mortality, myocardial infarction, any revascularisation, stroke
Patient oriented composite endpoint | 24 months
  Composite of all-cause mortality, myocardial infarction, any revascularisation, stroke
Patient oriented composite endpoint | 36 months
  Composite of all-cause mortality, myocardial infarction, any revascularisation, stroke
Patient oriented composite endpoint | 48 months
  Composite of all-cause mortality, myocardial infarction, any revascularisation, stroke
Patient oriented composite endpoint | 60 months
  Composite of all-cause mortality, myocardial infarction, any revascularisation, stroke
All-cause mortality | 1 month
  Death of any cause including cardiac deaths and non-natural causes of death
All-cause mortality | 12 months
  Death of any cause including cardiac deaths and non-natural causes of death
All-cause mortality | 24 months
  Death of any cause including cardiac deaths and non-natural causes of death
All-cause mortality | 36 months
  Death of any cause including cardiac deaths and non-natural causes of death
All-cause mortality | 48 months
  Death of any cause including cardiac deaths and non-natural causes of death
All-cause mortality | 60 months
  Death of any cause including cardiac deaths and non-natural causes of death
All-cause mortality | 120 months
  Death of any cause including cardiac deaths and non-natural causes of death
Cardiac death | 1 month
  Death due to cardiac causes or if death is not clearly attributable to other non-cardiac causes
Cardiac death | 12 months
  Death due to cardiac causes or if death is not clearly attributable to other non-cardiac causes
Cardiac death | 24 months
  Death due to cardiac causes or if death is not clearly attributable to other non-cardiac causes
Cardiac death | 36 months
  Death due to cardiac causes or if death is not clearly attributable to other non-cardiac causes
Cardiac death | 48 months
  Death due to cardiac causes or if death is not clearly attributable to other non-cardiac causes
Cardiac death | 60 months
  Death due to cardiac causes or if death is not clearly attributable to other non-cardiac causes
Myocardial infarction | 1 month
  Procedure and non-procedure related myocardial infarction
Myocardial infarction | 12 months
  Procedure and non-procedure related myocardial infarction
Myocardial infarction | 24 months
  Procedure and non-procedure related myocardial infarction
Myocardial infarction | 36 months
  Procedure and non-procedure related myocardial infarction
Myocardial infarction | 48 months
  Procedure and non-procedure related myocardial infarction
Myocardial infarction | 60 months
  Procedure and non-procedure related myocardial infarction
Stent Thrombosis | 1 month
  Definite, possible or probable
Stent Thrombosis | 12 months
  Definite, possible or probable
Stent Thrombosis | 24 months
  Definite, possible or probable
Stent Thrombosis | 36 months
  Definite, possible or probable
Stent Thrombosis | 48 months
  Definite, possible or probable
Stent Thrombosis | 60 months
  Definite, possible or probable
Target lesion myocardial infarction | 1 month
  Myocardial infarction related to an index treated lesion
Target lesion myocardial infarction | 12 months
  Myocardial infarction related to an index treated lesion
Target lesion myocardial infarction | 24 months
  Myocardial infarction related to an index treated lesion
Target lesion myocardial infarction | 36 months
  Myocardial infarction related to an index treated lesion
Target lesion myocardial infarction | 48 months
  Myocardial infarction related to an index treated lesion
Target lesion myocardial infarction | 60 months
  Myocardial infarction related to an index treated lesion
Target lesion revascularisation | 1 month
  Coronary artery bypass grafting or PCI of target lesion
Target lesion revascularisation | 12 months
  Coronary artery bypass grafting or PCI of target lesion
Target lesion revascularisation | 24 months
  Coronary artery bypass grafting or PCI of target lesion
Target lesion revascularisation | 36 months
  Coronary artery bypass grafting or PCI of target lesion
Target lesion revascularisation | 48 months
  Coronary artery bypass grafting or PCI of target lesion
Target lesion revascularisation | 60 months
  Coronary artery bypass grafting or PCI of target lesion
Target bifurcation myocardial infarction | 1 month
  Myocardial infarction related to the index bifurcation
Target bifurcation myocardial infarction | 12 months
  Myocardial infarction related to the index bifurcation
Target bifurcation myocardial infarction | 24 months
  Myocardial infarction related to the index bifurcation
Target bifurcation myocardial infarction | 36 months
  Myocardial infarction related to the index bifurcation
Target bifurcation myocardial infarction | 48 months
  Myocardial infarction related to the index bifurcation
Target bifurcation myocardial infarction | 60 months
  Myocardial infarction related to the index bifurcation
Target bifurcation revascularisation | 1 month
  Coronary artery bypass grafting or PCI of target bifurcation
Target bifurcation revascularisation | 12 months
  Coronary artery bypass grafting or PCI of target bifurcation
Target bifurcation revascularisation | 24 months
  Coronary artery bypass grafting or PCI of target bifurcation
Target bifurcation revascularisation | 36 months
  Coronary artery bypass grafting or PCI of target bifurcation
Target bifurcation revascularisation | 48 months
  Coronary artery bypass grafting or PCI of target bifurcation
Target bifurcation revascularisation | 60 months
  Coronary artery bypass grafting or PCI of target bifurcation
Target vessel revascularisation | 1 month
  Coronary artery bypass grafting or PCI of target vessel
Target vessel revascularisation | 12 months
  Coronary artery bypass grafting or PCI of target vessel
Target vessel revascularisation | 24 months
  Coronary artery bypass grafting or PCI of target vessel
Target vessel revascularisation | 36 months
  Coronary artery bypass grafting or PCI of target vessel
Target vessel revascularisation | 48 months
  Coronary artery bypass grafting or PCI of target vessel
Target vessel revascularisation | 60 months
  Coronary artery bypass grafting or PCI of target vessel
Any revascularisation | 1 month
  Any repeat revascularization except staged revascularization planned during the index procedure
Any revascularisation | 12 months
  Any repeat revascularization except staged revascularization planned during the index procedure
Any revascularisation | 24 months
  Any repeat revascularization except staged revascularization planned during the index procedure
Any revascularisation | 36 months
  Any repeat revascularization except staged revascularization planned during the index procedure
Any revascularisation | 48 months
  Any repeat revascularization except staged revascularization planned during the index procedure
Any revascularisation | 60 months
  Any repeat revascularization except staged revascularization planned during the index procedure
CCS angina class | 1 month
  Canadian Cardiovascular Society (CCS) grading of angina pectoris
CCS angina class | 12 months
  Canadian Cardiovascular Society (CCS) grading of angina pectoris
CCS angina class | 24 months
  Canadian Cardiovascular Society (CCS) grading of angina pectoris
CCS angina class | 36 months
  Canadian Cardiovascular Society (CCS) grading of angina pectoris
CCS angina class | 48 months
  Canadian Cardiovascular Society (CCS) grading of angina pectoris
CCS angina class | 60 months
  Canadian Cardiovascular Society (CCS) grading of angina pectoris
Post-PCI minimal lumen diameter in the stented proximal main vessel segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in the stented proximal main vessel segment
Post-PCI minimal lumen diameter in the stented distal main vessel segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in the stented distal main vessel segment
Post-PCI minimal lumen diameter in the treated side branch vessel segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in the treated (stent or balloon) side branch vessel segment
Post-PCI minimal lumen diameter in the proximal main vessel edge segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in the proximal main vessel edge segment (within 5 mm from the stent)
Post-PCI minimal lumen diameter in the distal main vessel edge segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in the distal main vessel edge segment (within 5 mm from the stent)
Post-PCI minimal lumen diameter in the side branch vessel edge segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in the side branch vessel edge segment (within 5 mm from stent or balloon)
Post-PCI minimal lumen diameter in the stented bifurcation core segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in the stented bifurcation core segment
Post-PCI minimal lumen diameter in the stented distal main vessel ostium segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in the stented distal main vessel ostium segment
Post-PCI minimal lumen diameter in the treated side branch vessel ostium segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in the treated side branch vessel ostium segment
Post-PCI diameter stenosis in the stented proximal main vessel segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in the stented proximal main vessel segment
Post-PCI diameter stenosis in the stented distal main vessel segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in the stented distal main vessel segment
Post-PCI diameter stenosis in the treated side branch vessel segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in the treated (stent or balloon) side branch vessel segment
Post-PCI diameter stenosis in the proximal main vessel edge segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in the proximal main vessel edge segment (within 5 mm from the stent)
Post-PCI diameter stenosis in the distal main vessel edge segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in the distal main vessel edge segment (within 5 mm from the stent)
Post-PCI diameter stenosis in the side branch vessel edge segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in the side branch vessel edge segment (within 5 mm from stent or balloon)
Post-PCI diameter stenosis in the stented bifurcation core segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in the stented bifurcation core segment
Post-PCI diameter stenosis in the stented distal main vessel ostium segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in the stented distal main vessel ostium segment
Post-PCI diameter stenosis in the treated side branch ostium segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in the treated side branch ostium segment
Post-PCI minimal lumen diameter in non-bifurcation target stented segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in non-bifurcation target stented segment
Post-PCI minimal lumen diameter in non-bifurcation target proximal edge segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in non-bifurcation target proximal edge segment (within 5mm fra stent)
Post-PCI minimal lumen diameter in non-bifurcation target distal edge segment | 1 day
  Post-PCI minimal lumen diameter by quantitative coronary analysis (QCA) in non-bifurcation target distal edge segment (within 5mm fra stent)
Post-PCI diameter stenosis in non-bifurcation target stented segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in non-bifurcation target stented segment
Post-PCI diameter stenosis in non-bifurcation target proximal edge segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in non-bifurcation target proximal edge segment
Post-PCI diameter stenosis in non-bifurcation target distal edge segment | 1 day
  Post-PCI diameter stenosis by quantitative coronary analysis (QCA) in non-bifurcation target distal edge segment

CONTACTS AND LOCATIONS:
Overall Officials: Evald H Christiansen, MD, PhD, Study Chair — Aarhus University Hospital, Denmark
Locations (38):
- Belgium (2):
  - Ziekenhuis Oost-Limburg (ZOL) Genk, Genk
  - Leuven University Hospital, Leuven
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital Skejby, Aarhus N
  - Gentofte Hospital, Gentofte Municipality
  - Rigshospitalet, København Ø
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde Sygehus, Roskilde
- Estonia Medical Centre, Tallinn, Estonia
- Tampere University Hospital, Tampere, Finland
- Germany (4):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Cardiologicum Hamburg, Hamburg
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
- University Hospital Galway, Galway, Ireland
- Italy (2):
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara, Cona
  - Gemelli General Hospital, Catholic University of the Sacred Heart, Rome
- Latvia Centre of Cardiology, Riga, Latvia
- Netherlands (3):
  - Northwest Hospital Alkmaar, Alkmaar
  - VU University Medical Center (VUMC), Amsterdam
  - St Antonius Ziekenhuis, Nieuwegein
- Norway (5):
  - Hospital of Southern Norway, Arendal, Arendal
  - Haukeland University Hospital, Bergen, Bergen
  - Oslo University Hospital, Rikshospitalet, Oslo
  - Oslo University Hospital - Ullevål, Oslo
  - Trondheim University Hospital, Trondheim
- Medical University of Warsaw, Warsaw, Poland
- Sweden (4):
  - Karolinska University Hospital Huddinge, Huddinge, Stockholm County
  - Sahlgrenska University Hospital, Gothenburg
  - Örebro University Hospital, Örebro
  - Södersjukhuset, Stockholm
- United Kingdom (7):
  - Belfast Health and Social Care Trust, Belfast
  - Royal Bournemouth Hospital, Bournemouth
  - Sussex Cardiac Centre, Brighton
  - Golden Jubilee Hospital, Glasgow
  - St George's Hospital, London
  - University Hospital South Manchester, Wythenshawe Hospital, Manchester
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Undecided
Is decided after primary endpoint assessment and requires regulatory approval

REFERENCES:
- [Derived] Holm NR, Andreasen LD, Neghabat O, Laanmets P, Kumsars I, Bennett J, Olsen NT, Odenstedt J, Hoffmann P, Dens J, Chowdhary S, O'Kane P, Bulow Rasmussen SH, Heigert M, Havndrup O, Van Kuijk JP, Biscaglia S, Mogensen LJH, Henareh L, Burzotta F, H Eek C, Mylotte D, Llinas MS, Koltowski L, Knaapen P, Calic S, Witt N, Santos-Pardo I, Watkins S, Lonborg J, Kristensen AT, Jensen LO, Calais F, Cockburn J, McNeice A, Kajander OA, Heestermans T, Kische S, Eftekhari A, Spratt JC, Christiansen EH; OCTOBER Trial Group. OCT or Angiography Guidance for PCI in Complex Bifurcation Lesions. N Engl J Med. 2023 Oct 19;389(16):1477-1487. doi: 10.1056/NEJMoa2307770. Epub 2023 Aug 27. PMID 37634149
- [Derived] Holm NR, Andreasen LN, Walsh S, Kajander OA, Witt N, Eek C, Knaapen P, Koltowski L, Gutierrez-Chico JL, Burzotta F, Kockman J, Ormiston J, Santos-Pardo I, Laanmets P, Mylotte D, Madsen M, Hjort J, Kumsars I, Ramunddal T, Christiansen EH. Rational and design of the European randomized Optical Coherence Tomography Optimized Bifurcation Event Reduction Trial (OCTOBER). Am Heart J. 2018 Nov;205:97-109. doi: 10.1016/j.ahj.2018.08.003. Epub 2018 Aug 16. PMID 30205242